CLINICAL TRIAL: NCT01334333
Title: Comparison of Medication Adherence Between Once Daily Tacrolimus (Advagraf®) and Twice Daily Tacrolimus (Prograf®) Administration in Stable Renal Transplant Recipients - a Randomized Study
Brief Title: Comparison of Medication Adherence Between Once and Twice Daily Tacrolimus in Stable Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Simon Fraser University (Other); Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H11-00446
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Renal Disease; Renal Transplant
Keywords: kidney transplant; tacrolimus; medication adherence; depression; neuropsychological; cognition; Self-efficacy; everyday problem solving
MeSH Terms: conditions — Kidney Diseases; Medication Adherence; Depression | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prograf® (Active Comparator): Prograf® is a twice daily formulation of tacrolimus
  Interventions: Drug: Tacrolimus - Prograf® twice daily formulation
- Advagraf® (Experimental): Advagraf® is a once daily formulation of tacrolimus
  Interventions: Drug: Tacrolimus - Advagraf® once daily formulation

INTERVENTIONS:
Drug: Tacrolimus - Prograf® twice daily formulation — twice daily, dosage will be as determined by best treatment for each participant, duration of study period will be 4 months for each participant
  Other Names: Prograf®
  Arms: Prograf®
Drug: Tacrolimus - Advagraf® once daily formulation — once daily, dosage will be as determined by best treatment for each participant, duration of study period will be 4 months for each participant
  Other Names: Advagraf®
  Arms: Advagraf®

SUMMARY:
A critical aspect of real-world functioning following kidney transplantation involves how adherent individuals are to their medication regimens. Regardless of the possible dangers of failing to adhere to anti-rejection medications, such as increased graft rejection, studies have reported rates of non-adherence at almost 50% following renal transplant.

The Cognitive Aging Laboratory under the direction of Dr. Wendy Thornton, at Simon Fraser University, has previously identified relationships between several potentially important cognitive and psychosocial variables, and self-reported medication adherence in renal transplant recipients, including depressive symptoms, as well as everyday and traditional cognitive functioning [4]. The possibility that changes in dosing regimens for a given medication may have an additional impact on medication adherence presents an important issue worth further exploration.

The current study will allow for more thorough delineation of the roles of psychosocial and cognitive predictors of adherence with state-of-the-art monitoring techniques. In addition, the investigators will assess whether different dosing formulations of tacrolimus impact adherence behaviors in renal transplant recipients.

The proposed research has two primary aims to examine:

1. To examine the role of cognitive and psychosocial variables in predicting medication adherence in renal transplant recipients.
2. To examine whether different formulations of tacrolimus (once per day dosing versus twice per day dosing) will impact medication adherence in renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* a minimum of one year post renal transplant with a successful kidney graft and stable renal function (estimated glomerular filtration rate [GFR (glomerular filtration rate)] above 25 ml/minute per 1.73 m2).
* currently prescribed tacrolimus
* able to swallow pills
* a minimum of grade six education
* fluent in the English language.

Exclusion Criteria:

* refusal to or inability to give written informed consent.
* any visual, hearing or other sensory/motor impairments which may interfere with the testing procedures.
* have had a stroke determined to be of significant severity
* have had a head injury determined to be of significant severity
* have a current psychiatric diagnosis determined to be of significant severity
* have the presence of an acute illness (e.g., metastatic cancer), neurological disease, and other major organ failure (e.g., end stage liver disease)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-11-11 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
electronic monitor of medication taking | 4 months
  electronic bottle tops will be used to monitor medication adherence using MEMS (medication event monitoring system) Caps technology for a period of 4 months.

SECONDARY OUTCOMES:
blood levels of medication | 4 months
  blood levels of tacrolimus will be monitored throughout the study.
self-reported medication adherence | 4 months
  self-report medication adherence questionnaires will also be used to assess medication adherence.
pharmacy refill data | 4 months
  pharmacy refill data from the hospital pharmacy where all participants receive their medications will also be examined to determine medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: R. Jean Shapiro, M.D., Principal Investigator — University of British Columbia; Wendy Loken Thornton, Ph.D., Principal Investigator — Simon Fraser University; Nilufar Partovi, Pharm.D., Principal Investigator — University of British Columbia; Theone SE Paterson, M.A., Principal Investigator — Simon Fraser University
Locations (1):
- Solid Organ Transplant Clinic, Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- [Derived] Paterson TSE, Demian M, Shapiro RJ, Loken Thornton W. Impact of Once- Versus Twice-Daily Tacrolimus Dosing on Medication Adherence in Stable Renal Transplant Recipients: A Canadian Single-Center Randomized Controlled Trial. Can J Kidney Health Dis. 2019 Aug 17;6:2054358119867993. doi: 10.1177/2054358119867993. eCollection 2019. PMID 31452902